CLINICAL TRIAL: NCT00761046
Title: Retrospective Study on Cenos Stem With BoneMaster HA
Status: Withdrawn | Type: Observational
Why Stopped: No data have been obtained at all in this time.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: BMET DE 02
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Retrospective data collection of the CENOS implant comparing with and without BoneMaster HA coatings.

DETAILED DESCRIPTION:
Not applicable as study was withdrawn

ELIGIBILITY:
Patients Who Received CENOS prosthesis for Intended Uses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients Who Received CENOS prosthesis for Intended Uses
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-10

PRIMARY OUTCOMES:
Complication Rate